CLINICAL TRIAL: NCT04698798
Title: Skeletal Muscle Wasting in SARS-CoV-2 Infected ICU (Intensive Care Unit) Patients
Brief Title: Skeletal Muscle Wasting in SARS-CoV-2
Acronym: SMW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Frank Vandenabeele, Principal Investigator, Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SMW-CoV-2
Record Dates: First submitted 2021-01-04; First posted 2021-01-07 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Cachexia; Muscle Loss; Muscle Wasting; Muscle Atrophy; Critical Illness
MeSH Terms: conditions — Cachexia; Muscular Atrophy; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Skeletal muscle wasting (Experimental): investigating acute skeletal muscle wasting in patients infected with SARS-CoV-2 and admitted to the ICU
  Interventions: Procedure: Muscle Biopsy

INTERVENTIONS:
Procedure: Muscle Biopsy — Patients will be treated for SARS-CoV-2 symptoms on the intensive care unit. During this treatment two muscle biopsies will be obtained with an interval of seven days between them.

SUMMARY:
The SARS-CoV-2 pandemic causes a major burden on patient and staff admitted/working on the intensive care unit (ICU). Short, and especially long admission on the ICU causes major reductions in skeletal muscle mass (3-4% a day) and strength. Since it is now possible to reduce mortality on the ICU, short and long-term morbidity should be considered another principal endpoint after SARS-CoV-2 infection. Cachexia is defined as 'a complex metabolic syndrome associated with underlying illness and characterized by loss of muscle mass'. Its clinical features are weight loss, low albumin, anorexia, increased muscle protein breakdown and inflammation. There is strong evidence that cachexia develops rapidly in patients hospitalized for SARS-CoV-2 infection, especially on the ICU. Several mechanisms are believed to induce cachexia in SARS-CoV-2. Firstly, the virus can interact with muscle cells, by binding to the angiotensin converting enzyme 2 (ACE-2). In vitro studies have shown the virus can cause myofibrillar fragmentation into individual sarcomeres, in addition to loss of nuclear DNA in cardiomyocytes. Similar results were found during autopsies. On a cellular level, nothing is known about the effects of SARS-CoV-2 infection on skeletal muscle cells. However, up to 19.4% of patients present with myalgia and elevated levels of creatine kinases (>200U/l), suggesting skeletal muscle injury. Moreover, patients with SARS-CoV-2 infection are shown to have elevated levels of C-reactive protein and other inflammatory cytokines which can all affect skeletal muscles. The above mentioned factors are not the only mediators by which skeletal muscle mass might be affected in SARS-CoV-2. There are other known factors to affect skeletal muscle mass on the ICU, i.e. immobilization and mechanical ventilation, dietary intake (anorexia) and inflammatory cytokines. SARS-CoV-2 infection in combination with bed rest and mechanical ventilation can lead to severe muscle wasting and functional decline resulting in long-term morbidity.

Until know there are no studies investigating acute skeletal muscle wasting in patients infected with SARS-CoV-2 and admitted to the ICU. As a result, there is a need of more in-depth understanding the effects of SARS-CoV-2 infection on muscle wasting. An optimal characterization of these effects may lead to improvement in morbidity and even mortality in the short and long term by the establishment of evidence-based rehabilitation programs for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* SARS-CoV-2 infection
* Expected stay to ICU of > 7 days

Exclusion Criteria:

* Spinal cord injury
* Chronic use of corticosteroids before hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2021-04-03 (Actual); Study Completion 2021-04-03 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle biopsy | baseline
  A muscle biopsy of the m. vastus lateralis will be obtained at T0, after admission on ICU to evaluate the effects of SARS-CoV-2 infection and ICU admission on skeletal muscle fiber characteristics Muscle biopsy samples will be obtained using a minimally invasive (Bard® Mission® Core Biopsy Instrument (14G 10mm needle)) biopsy technique, under local anaesthesia
Skeletal muscle biopsy | Day 7
  A muscle biopsy of the m. vastus lateralis will be obtained at T4, after admission on ICU to evaluate the effects of SARS-CoV-2 infection and ICU admission on skeletal muscle fiber characteristics Muscle biopsy samples will be obtained using a minimally invasive (Bard® Mission® Core Biopsy Instrument (14G 10mm needle)) biopsy technique, under local anaesthesia
Electrophysiological test | Baseline
  Electrophysiological test will be performed at T0 and T1. For nerve conduction studies, one standard motor and one sensory nerve will be evaluated in both upper and lower limbs unilaterally. We define reduced CMAP and SNAP when below the lower limit of normal in both nerves of both limbs. Needle electromyography in rest will be performed unilaterally in one standard proximal and distal muscle in both upper and lower limbs. Abundant SEA was defined as the presence of sustained fibrillation potentials and/or positive sharp waves in at least two muscles of at least two limbs.
Electrophysiological test | Day 7
  Electrophysiological test will be performed at T0 and T1. For nerve conduction studies, one standard motor and one sensory nerve will be evaluated in both upper and lower limbs unilaterally. We define reduced CMAP and SNAP when below the lower limit of normal in both nerves of both limbs. Needle electromyography in rest will be performed unilaterally in one standard proximal and distal muscle in both upper and lower limbs. Abundant SEA was defined as the presence of sustained fibrillation potentials and/or positive sharp waves in at least two muscles of at least two limbs.

SECONDARY OUTCOMES:
Skeletal muscle biopsy | Baseline
  Secondary outcome from the biopsy samples will focus on muscle fiber typing, muscle fiber type-specific CSA, muscle fiber type-specific myonuclear content, muscle fiber type-specific satellite cell content, muscle fiber type-specific capillaries, muscle resident/infiltrating macrophages and others using immunohistochemical stainings. RNA analyses will be done by RT-PCR, and protein analyses by Western Blot for different markers related to oxidative stress, protein synthesis, protein degradation. Myofibrillar damage and viral cell infiltrates and other possible structural changes will be analysed using transmission electron microscopy.
Skeletal muscle biopsy | Day 7
  Secondary outcome from the biopsy samples will focus on muscle fiber typing, muscle fiber type-specific CSA, muscle fiber type-specific myonuclear content, muscle fiber type-specific satellite cell content, muscle fiber type-specific capillaries, muscle resident/infiltrating macrophages and others using immunohistochemical stainings. RNA analyses will be done by RT-PCR, and protein analyses by Western Blot for different markers related to oxidative stress, protein synthesis, protein degradation. Myofibrillar damage and viral cell infiltrates and other possible structural changes will be analysed using transmission electron microscopy.
Blood sample analyses | daily between baseline and day 7
  Standard blood work will be queried during the trial period. We will especially focus on blood marker for muscle damage (such as CK, LDH…) and inflammation (CRP, WBC…).
Mechanical ventilation and oxygen therapy | daily between baseline and day 7
  the modality of oxygen therapy or mechanical ventilation will be monitored each day the patient is in the trial.
Dietary intake | daily between baseline and day 7
  Dietary intake will be monitored every day the patient is within the trial. It will be monitored if the patient receives standard feeding, total parenteral feeding or others. Description: the modality of oxygen therapy or mechanical ventilation will be monitored each day the patient is in the trial.
concommitted medication | daily between baseline and day 7
  All medication that the patients receive will be monitored during the period they participate within the trial.
APACHE II score | Baseline
  Acute Physiology and Chronic Health Evaluation II (APACHE II) is a severity-of-disease classification system. An integer score from 0 to 71 will be computed based on several measurements; higher scores correspond to more severe disease and a higher risk of death.
APACHE II score | day 7
  Acute Physiology and Chronic Health Evaluation II (APACHE II) is a severity-of-disease classification system. An integer score from 0 to 71 will be computed based on several measurements; higher scores correspond to more severe disease and a higher risk of death.
Comorbidities | baseline
  All comorbidities will be obtained from the patients medical file.
Duration from hospital admission to ICU admission | baseline
  The duration from hospital admission to ICU admission will be noted at T0. This will be done because the amount of days patients are already in the hospital could influence the amount of skeletal muscle atrophy in the ICU.
Symptoms of disease onset and myalgia | baseline
  symptoms of disease onset (fever, cough, anorexia, throat pain, abdominal pain, myalgia, neurological symptoms) will be noted at T0.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Vandenabeele, prof. dr., Principal Investigator — Hasselt University; Sjoerd stevens, drs., Study Chair — Hasselt University
Locations (1):
- Jessa Ziekenhuis, Hasselt, Belgium